CLINICAL TRIAL: NCT03671915
Title: An Open-label, Three-center, Randomized, Two-session, Crossover Study, to Assess 4 Days Inpatient, and 6-week Follow-up Home Study Phase Under Remote Monitoring at Only French Centers, the Efficacy and the Safety of the Diabeloop Closed-loop Glucose Control Compared With Sensor-augmented Pump Therapy, in Young Children With Type 1 Diabetes.
Brief Title: Diabeloop for Kids
Acronym: DBL4K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02078-47
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Closed Loop; Diabetes Mellitus, Type 1; Young Children (6 to 12 Years Old )
Keywords: artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring; Telemedicine

STUDY DESIGN:
Intervention Model Description: Closed loop vs. Open loop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual System (Open-loop) (Active Comparator): In open loop: sensor-augmented pump (SAP) therapy using standard insulin pump setting combined with the six-generation glucose sensor (Dexcom G6).
  Interventions: Device: Continuous Glucose Monitoring; Device: External Insulin Pump
- DIABELOOP System (Closed-loop) (Experimental): In the closed loop: Diabeloop software (an MPC-based glucose control algorithm) running on handset associated with the six-generation glucose sensor (Dexcom G6) and Kaleïdo insulin pump.
  A remote monitoring system managed by specialized nurse on behalf diabetologist, is provided in closed-loop session.
  Interventions: Device: Continuous Glucose Monitoring; Device: External Insulin Pump; Device: Diabeloop Software (Model predictive control); Other: Remote monitoring (Telemedicine)

INTERVENTIONS:
Device: Continuous Glucose Monitoring — collection of glucose data
Device: External Insulin Pump — Insulin delivery
Device: Diabeloop Software (Model predictive control) — Diabeloop software embeds a regulation algorithm to automatically regulate the patient's glycaemia. It takes as input glycaemia value received every 5 minutes from the CGM and patient inputs related to meals and physical activities and it calculates the amount of insulin to be delivered. It sends this information to the pump that automatically delivers this quantity.
  Arms: DIABELOOP System (Closed-loop)
Other: Remote monitoring (Telemedicine) — Remote follow up by care health providers team
  Arms: DIABELOOP System (Closed-loop)

SUMMARY:
An open-label, three-center, randomized, two-session, 4 days inpatient and 6-week follow-up home study phase, crossover study comparing Diabeloop closed-loop (CL) system and sensor-augmented pump (SAP) therapy.

The follow-up home study phase will be done only in French centers for a sub study. During this session, patient wearing the closed-loop system will benefit of a 24h/24, 7 d/7, remote monitoring follow-up by specialized nurses, under supervision of a diabetologist. A visualization of glucose CGM curves, insulin delivery, meal and physical activity announcements will be available online through secured website, and the system will send automated message in case of predetermined situations as persistent too high or too low Blood Glucose (BG). Custom settings will be possible by the nurses during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Prepubescent children (Gender: both) aged between 6 to 12 years old (Tanner stage 1) at time of screening
* Type 1 diabetes as defined by WHO for at least 1 year or confirmed C peptide negative
* An insulin pump user for at least 3 months.
* Subject having a Glycosylated hemoglobin (HbA1c) blood value < 9% at time of screening visit-based on analysis from local laboratory within 3 months.
* Subject having a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units.
* Subject and his parent/guardian willing to spend 3-overnight in hospital.
* Subject willing to wear the system continuously throughout the study
* Subjects and his parent/guardian must be able to speak and be literate in French or Flemish as verified by the investigator

Exclusion Criteria:

* Children who are in pubertal stage
* Subject has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening: - Medical assistance (i.e. Paramedics, Emergency Room (ER) or Hospitalization) - Coma - Seizures
* Subject having sever DKA in the 6 months prior to screening visit.
* Known or suspected allergy against insulin
* Any other physical or psychological disease, or medication likely to interfere with the conduct of the study and interpretation of the study results as judged by the investigator.
* Subject is unable to tolerate tape adhesive around the sensor or pump placements
* Subject has a cardiovascular condition which the investigator determines should exclude the subject, i.e. ventricular rhythm disturbance, hypertrophic cardiomyopathy
* Subject having took any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
The time spent of the glucose level drop in below 70 mg/dl over the 72-h, as recorded by continuous subcutaneous glucose monitoring (CGM). | 72 hours
  Measurement of glucose by CGM

SECONDARY OUTCOMES:
Sensor mean glucose | 72 hours, in the overnight (defined as 23:00 to 07:00) and 6 weeks (home study phase)
  Sensor mean glucose over the 72-h, in the overnight (defined as 23:00 to 07:00) and during the home study phase for the French centers, in closed-loop and open-loop session
Coefficient of variation (SD/Mean %) | 72 hours
Standard deviation (SD mg/dl) of the glucose rate of change as recorded by the CGM | 72 hours
  Measurement of glucose by CGM
Low Blood Glucose Index (LBGI) and high blood glucose Index (HBGI) | 72 hours and 6 weeks (home study phase)
  Measurement of glucose by CGM
Percentage of sensor time in glucose range 70-140 mg/dl | 72 hours and 6 weeks (home study phase)
  Measurement of glucose by CGM
Percentage time in glucose levels in the widened target range 70-180 mg/dl | 72 hours and 6 weeks (home study phase)
  Measurement of glucose by CGM
Fasting blood glucose, mg/dl (mmol/L) | 72 hours and 6 weeks
Sensor time spent in glucose levels below 54 mg/dl, 60 mg/dl | 72 hours
  Measurement of glucose by CGM
Sensor time spent in glucose levels below 54 mg/dl, 60 mg/dl, and 70 mg/dl | 72 hours, in the overnight (defined as 23:00 to 07:00) and 6 weeks (home study phase)
  Measurement of glucose by CGM
Number of severe Hyperglycemic events as well as the number of subjects experiencing sever hypoglycemia | 72 hours and 6 weeks (home study phase)
  Measurement of glucose by CGM
Time spent in glucose levels above 180 mg/dl, 250 mg/dl, 300 mg/dl | 72 hours, in the overnight (defined as 23:00 to 07:00) and 6 weeks (home study phase)
  Measurement of glucose by CGM
Severe Diabetic Ketoacidosis (DKA) events | 72 hours and 6 weeks (home study phase)
  Subjects will be asked to measure blood urine ketone levels on waking in the morning if their finger-stick glucose is above 200 mg/l, as part of the safety evaluation for hyperglycemia.
Percentage of time closed-loop active | 72 hours and 6 weeks (home study phase)
Total daily dose of insulin | 72 hours and 6 weeks (home study phase)
  Total basal and bolus by 24h
Subject's perception in terms of life-style change, satisfaction and diabetes management | 72 hours and 6 weeks (home study phase)
  Subject's perception in terms of life-style change, satisfaction and diabetes management as evaluated by PedsQL, DTQ, DTSQ and AP acceptance questionnaire.

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- France (2):
  - Necker Enfants Malades Hospital, Paris
  - Toulouse University Hospital Center, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benhamou PY, Adenis A, Tourki Y, Pou S, Madrolle S, Franc S, Kariyawasam D, Beltrand J, Klonoff DC, Charpentier G. Efficacy of a Hybrid Closed-Loop Solution in Patients With Excessive Time in Hypoglycaemia: A Post Hoc Analysis of Trials With DBLG1 System. J Diabetes Sci Technol. 2024 Mar;18(2):372-379. doi: 10.1177/19322968221128565. Epub 2022 Sep 29. PMID 36172702
- [Derived] Kariyawasam D, Morin C, Casteels K, Le Tallec C, Sfez A, Godot C, Huneker E, Garrec N, Benhamou PY, Polak M, Charpentier G, Franc S, Beltrand J. Hybrid closed-loop insulin delivery versus sensor-augmented pump therapy in children aged 6-12 years: a randomised, controlled, cross-over, non-inferiority trial. Lancet Digit Health. 2022 Mar;4(3):e158-e168. doi: 10.1016/S2589-7500(21)00271-5. PMID 35216750